CLINICAL TRIAL: NCT05936775
Title: Assessment of Osseointegration Properties of Nano-Hydroxy Apatite Coated Titanium Implant Versus Sandblasted Large Thread Acid Etched Implants in Posterior Maxilla. A Randomized Clinical Trial
Brief Title: Assessment of Osseointegration Properties of Nano-Hydroxy Apatite Coated Titanium Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Mohamed Hamdy Mahmoud Ismail, Lecturer, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2023-06-22; First posted 2023-07-10 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Implant Site Reaction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nano-hydroxy apatite arm (Experimental): in this groups patients will receive nano-hydroxy apatite coated titanium implants
  Interventions: Other: nano-hydroxy apatite coated titanium implants
- SLA arm (Active Comparator): in this group patients will receive sandblasted large thread acid etched titanium implants
  Interventions: Other: sandblasted large acid itched coated titanium implant

INTERVENTIONS:
Other: nano-hydroxy apatite coated titanium implants — titanium implants with surface treatment of nano-hydroxy apatite
  Arms: Nano-hydroxy apatite arm
Other: sandblasted large acid itched coated titanium implant — titanium implants with SLA surface treatment
  Arms: SLA arm

SUMMARY:
the purpose of this trial is to evaluate the osseointegration properties of nano-hydroxy apatite coated titanium implants in posterior maxilla. 30 patients will be included in this trial divided into two groups, control and intervention. Primary and secondary implant stability will be measured

ELIGIBILITY:
Inclusion Criteria:

1. Patients with missing at least one maxillary posterior tooth
2. Patients free from any systemic disease
3. Patients who approve to be included in the trial and sign the informed consent
4. Patients with no intra-bony defect.
5. Adults aged 18 years old and above

Exclusion Criteria:

1. Patients who are allergic to titanium
2. Heavy smoker patient
3. Patients receiving chemotherapy or radiotherapy
4. Patients who refused to be included in the trial

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Implant stability | immediately post-operative
  implant stability will be measured by radiofrequency analysis
Implant stability | 4 weeks post-operative
  implant stability will be measured by radiofrequency analysis
Implant stability | 6 weeks post-operative
  implant stability will be measured by radiofrequency analysis
Implant stability | 12 weeks post-operative
  implant stability will be measured by radiofrequency analysis

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Mahmoud, PhD, Principal Investigator — october university for modern science and arts faculty of dentistry
Locations (1):
- October University for Modern Sciences and Arts faulty of Dentistry, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No